CLINICAL TRIAL: NCT00675597
Title: A Pilot Study of Docetaxel (Taxotere), Vinorelbine, and Bevacizumab, as Adjuvant Chemotherapy for Patients With Resected Stage I-III Non-small Cell Lung Cancer
Brief Title: Docetaxel (Taxotere), Vinorelbine, and Bevacizumab, as Adjuvant Chemotherapy for Patients With Resected Stage I-III Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-178
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: Bevacizumab (Avastin); Taxotere (Docetaxel); Vinorelbine Tartrate (Navelbine); 07-178
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab; Docetaxel; Vinorelbine

ARMS (1):
- 1 (Experimental): Docetaxel (Taxotere), Vinorelbine, and Bevacizumab, as Adjuvant Chemotherapy for Patients with Resected Stage I-III Non-small Cell Lung Cancer
  Interventions: Drug: Bevacizumab (Avastin), Taxotere (Docetaxel), Vinorelbine Tartrate (Navelbine)

INTERVENTIONS:
Drug: Bevacizumab (Avastin), Taxotere (Docetaxel), Vinorelbine Tartrate (Navelbine) — Patients will be treated as follows: vinorelbine (45 mg/m2) + docetaxel (45 mg/m2) intravenously on day 1, followed by pegylated filgrastim 6mg subcutaneously on day 2, delivered every 2 weeks for 8 doses total. Patients who have already received one cycle of cisplatin-based adjuvant chemotherapy need only complete 3 cycles of vinorelbine+docetaxel for a total of 4 cycles of adjuvant chemotherapy. Patients who require post-operative radiation therapy (PORT) will begin PORT after completion of vinorelbine + docetaxel.

SUMMARY:
The purpose of this study is to determine whether a combination of the drugs docetaxel (Taxotere ® ), plus vinorelbine (Navelbine ® ), will result in fewer side effects than cisplatin chemotherapy, thereby improving delivery of chemotherapy in patients.

Another purpose of this study is to determine whether a third drug, bevacizumab (Avastin®), may be delivered safely with docetaxel plus vinorelbine in patients who are eligible to receive bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 2 weeks status post complete (R0) surgical resection of pathologically-proven NSCLC (stage IA-IIIB). Pathology review will be performed independently at MSKCC.
* Patients are eligible if they are unfit for cisplatin-based adjuvant chemotherapy based on specified clinical criteria (listed below).
* Allergy to cisplatin
* Baseline hearing loss (defined as any subjective baseline hearing deficit, even if it does not require a hearing aid or intervention, or interfere with activities of daily life (CTCAE grade > or equal to 2)
* Baseline renal insufficiency (defined as a creatinine clearance of < than or equal to 60 ml/min as calculated by the equation of Cockcroft and Gault using the patient's age, weight (kg), and serum creatinine (mg/dl).
* Performance status 70% on the Karnofsky scale.
* Congestive heart failure with New York Heart Association functional classification > or equal to II, characterized by fatigue, dyspnea or other symptoms which limit activities of daily life.
* Patient refuses to take cisplatin.
* Age > than or equal 18
* Performance Status Karnofsky > than or equal to 70%
* Peripheral neuropathy must be < than grade 1
* Hematologic (minimal values)
* Absolute neutrophil count > than or equal to 1,500/mm3
* Hemoglobin > than or equal to 8.0 g/dl
* Platelet count > than or equal to 100,000/mm3 Hepatic
* Total Bilirubin < than or equal to 1.5 x ULN AST or ALT and Alkaline Phosphatase must be within the range allowing for eligibility
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients being considered for treatment with bevacizumab must have a urine protein: creatinine (UPC) ratio < 1.0 at screening and an MRI of brain or CT brain with IV contrast showing no evidence of brain metastases within 3 months of study entry

Exclusion Criteria:

* > 16 weeks post-op
* Prior post-operative radiation
* > 1 cycle of prior adjuvant chemotherapy
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Women who are pregnant, or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Azzoli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel (Taxotere®) Plus Vinorelbine: Docetaxel (Taxotere®) plus Vinorelbine as Adjuvant Chemotherapy for Patients with Resected Stage I-III Non-small Cell Lung Cancer
Period: Overall Study
Arm/Group | Docetaxel (Taxotere®) Plus Vinorelbine
Started | 26
Completed | 23
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel (Taxotere®) Plus Vinorelbine
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 64.6 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: To Measure the Number of Cycles
Description: Cycle delivery is a surrogate for drug delivery. Both cycle delivery and drug delivery will be measured in this study. However, cycle delivery (up to 4 cycles) is the common way drug delivery is measured in the literature, and therefore cycle delivery has been chosen as the primary endpoint for this study.Two doses of both docetaxel plus vinorelbine, delivered over 4 weeks, constitutes one cycle. If either drug is discontinued, the subject will remain on study, however that patient will not get credit for completing subsequent cycles of therapy. If the dose of either drug is reduced, the subject will remain on study and get credit for subsequent cycles.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Docetaxel (Taxotere®) Plus Vinorelbine
Number analyzed (Participants) | 23
participants
  Completed 4 cycles | 20
  Unable to complete 4 cycles | 3

ADVERSE EVENTS:
Arm/Group | Docetaxel (Taxotere®) Plus Vinorelbine
Serious Adverse Events (participants affected / at risk) | 13/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (Taxotere®) Plus Vinorelbine (N=23)
Nausea (General disorders) | 1 (1)
Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1)
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 5 (6)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Inf norm ANC/gr1/2 neut-Catheter-related (Blood and lymphatic system disorders) | 1 (1)
Inf unknown ANC-Ungual(nails) (Infections and infestations) | 1 (1)
Infection, other (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Mucositis (func/sympt)- Oral cavity (General disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3)
Pain - Abdomen NOS (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (Taxotere®) Plus Vinorelbine (N=23)
Fatigue (General disorders) | 14 (45)
Neuropathy (Nervous system disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 4 (4)
ALT, SGPT (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (8)
Cough (General disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (15)
Fever (in the absence of neutropenia) (General disorders) | 2 (3)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 16 (16)
Hair loss/alopecia (scalp or body) (General disorders) | 9 (9)
Hemoglobin (Blood and lymphatic system disorders) | 14 (14)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 13 (13)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Mucositis (Clin exam)- Oral cavity (General disorders) | 8 (8)
Nail changes (Skin and subcutaneous tissue disorders) | 5 (5)
Nausea (General disorders) | 3 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14 (14)
Pain - Other (General disorders) | 4 (5)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (3)
Watery eye (epiphora, tearing) (Eye disorders) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes